CLINICAL TRIAL: NCT06911008
Title: Phase I Trial of SCD I: A First in Human Dose Regimen-Finding Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Activity of MTI-301 in Patients With Advanced Malignancy
Brief Title: MTI-301 for the Treatment of Metastatic or Unresectable and Refractory Solid Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210103; NCI-2025-01930 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-012791 (Other: Mayo Clinic Institutional Review Board); MC210103 (Other: Mayo Clinic); R44CA272064 (NIH)
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (MTI-301) (Experimental): Patients receive MTI-301 PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, PET/CT, or MRI and collection of blood samples throughout the study, and undergo tissue sample collection at baseline and at disease progression.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Biological: SCD1 Inhibitor MTI-301

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo tissue and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Biological: SCD1 Inhibitor MTI-301 — Given PO
  Other Names: MTI-301; MTI301; MTI 301; Stearoyl-CoA Desaturase 1 Inhibitor MTI-301; SSI-4; SSI4; SSI 4; ); 2-{[4-(2-Chlorophenoxy)piperidine-1-carbonyl]amino}-N-methylpyridine-4-carboxamide

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of MTI-301 in treating patients with solid cancers that have spread from where they first started (primary site) to other places in the body (metastatic) or that cannot be removed by surgery (unresectable) and that have not responded to previous treatment (refractory). MTI-301 is a drug that inhibits an enzyme called SCD1. SCD1 is an enzyme that promotes tumor growth and spread and is upregulated in some cancer types. MTI-301 may disrupt the activity of SCD1, which may lead to reduced tumor growth and/or spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess and determine the maximum tolerated dose (MTD) for SCD1 inhibitor MTI-301 (MTI-301).

SECONDARY OBJECTIVES:

I. To determine the toxicity profile with MTI-301. II. To determine objective response rate (ORR), progression free survival (PFS) and duration of response (DOR).

CORRELATIVE RESEARCH:

I. To characterize the pharmacokinetic (PK) profile of MTI-301. II. To assess the levels of SCD1 substrates steric acid, palmitic acid and products oleic acid, palmitoleic acid at baseline, at progression, and at the end of study.

III. To assess immune regulator factors from blood at baseline, at progression, and at the end of study.

OUTLINE: This is a dose-escalation study of MTI-301.

Patients receive MTI-301 orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT), positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI) and collection of blood samples throughout the study, and undergo tissue sample collection at baseline and at disease progression.

After completion of study treatment, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically or cytologically confirmed solid tumor (cancer) that is metastatic or unresectable and who are refractory to or intolerant of existing, standard-of-care therapy(ies), known to provide clinical benefit for their condition.
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria or evaluable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2.
* Hemoglobin ≥ 9.0 g/dL (obtained ≤ 28 days prior to registration).
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained ≤ 28 days prior to registration).
* Platelet count ≥ 100,000/mm^3 (obtained ≤ 28 days prior to registration).
* Total bilirubin ≤ 1.5 x upper limit normal (ULN). Patients with Gilbert's syndrome: Total bilirubin ≤ 3 x ULN (obtained ≤ 28 days prior to registration).
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3 x ULN (≤ 5 x ULN for patients with liver involvement) (obtained ≤ 28 days prior to registration).
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy as determined by treating investigator (obtained ≤ 28 days prior to registration).
* Calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault formula (obtained ≤ 28 days prior to registration).
* Negative pregnancy test done ≤ 7 days prior to registration, for persons of childbearing potential only.

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Provide written informed consent.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Willingness to provide mandatory blood specimens for correlative research.
* Willingness to provide mandatory tissue specimens for correlative research.
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons who are of childbearing potential who are unwilling to employ adequate contraception.
  * NOTE: For the purpose of this guidance, methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods. Such methods include:

    * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation [Hormonal contraception may be susceptible to interaction with the investigational medicinal product (IMP), which may reduce the efficacy of the contraception method.]:

      * Oral
      * Intravaginal
      * Transdermal
    * Progestogen-only hormonal contraception associated with inhibition of ovulation (Hormonal contraception may be susceptible to interaction with the IMP, which may reduce the efficacy of the contraception method.):

      * Oral
      * Injectable
      * Implantable (Contraception methods that in the context of this guidance are considered to have low user dependency.)
    * Intrauterine device (IUD) (Contraception methods that in the context of this guidance are considered to have low user dependency)
    * Intrauterine hormone-releasing system (IUS) (Contraception methods that in the context of this guidance are considered to have low user dependency.)
    * Bilateral tubal occlusion (Contraception methods that in the context of this guidance are considered to have low user dependency.)
    * Vasectomised partner [Contraception methods that in the context of this guidance are considered to have low user dependency. Vasectomised partner is a highly effective birth control method provided that partner is the sole sexual partner of the women of childbearing potential (WOCBP) trial participant and that the vasectomised partner has received medical assessment of the surgical success.]
    * Sexual abstinence (In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.).
* Any of the following prior therapies:

  * Major surgery ≤ 3 weeks prior to registration
  * Chemotherapy ≤ 2 weeks prior to registration
  * Immunotherapy ≤ 3 weeks prior to registration
  * Radiation ≤ 2 weeks prior to registration.
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy, patients with hepatitis B and C on active treatment, or those with acute hepatitis B and C not currently on treatment.

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Clinically significant cardiac arrhythmia
  * Bleeding disorder
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
  * Any other conditions that would limit compliance with study requirements.
* History of myocardial infarction ≤ 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias.
* Other active malignancy ≤ 3 years prior to registration.

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix.
  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer.
* Unresolved toxicity from prior chemotherapy (subjects must be recovery to ≤ grade 1 toxicity from previous anticancer treatments or previous investigational agents).
* Receiving any other investigational agent or device ≤ 14 days prior to registration.
* Planning on receiving other medical, surgical, or radiological cancer treatments during the course of this study.
* Evidence of untreated fluid retention at the time of registration (including, for example, peripheral edema, pleural effusion, or ascites on physical or radiological examination) or history of severe capillary leak syndrome.
* Any other condition which the investigator believes would make participation in the study not acceptable.
* Subjects with any active and/or symptomatic brain metastases or active primary central nervous system (CNS) and subjects with carcinomatosis meningitis are excluded.

  * NOTE: History of brain metastases treated by surgery and/or radiotherapy provided neurologically stable and off steroids ≥ 4 weeks prior to registration are allowed.
* Grade 2 or greater neuropathy (excluding diagnosed carpal tunnel syndrome).
* Use of concomitant medication that are known to be inhibitors or substrates of major CYP enzymes, CYP2C9, CYP2c19, CYP3a4, CYP2D6, CYP1A2, CYP2B6 and CYP2C8 ≤ 14 days prior to registration.
* Use of concomitant medication that are known to be inhibitors or substrates of transporters ≤ 14 days prior to registration.
* Corrected QT (QTc) prolongation based on QTc interval prior to registration of ≥ 470 ms using the Fridericia's formula (QTcF).
* Confluent superficial keratitis, a cornea epithelial defect, a corneal ulcer or stromal opacity.
* Significant electrolyte imbalance.
* Significant uncontrolled congestive heart failure.
* Symptomatic uncontrolled cardiac arrhythmia.
* Genetic predisposition for long QT syndrome.
* Subjects who are receiving concomitant QT prolonging medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-04-09 (Estimated); Study Completion 2027-04-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 28 days (1 cycle)
  Will be defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients). DLT will be defined as an adverse event attributed as definitely, probably, or possibly related to MTI-301.
Incidence of adverse events | Up to 30 days after last dose of study treatment
  Will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized. Grade 3+ adverse events will be described and summarized in a similar fashion. This will provide an indication of the level of tolerance for this treatment combination.

SECONDARY OUTCOMES:
Objective response rate | Up to 6 cycles (1 cycle = 28 days)
  Will be defined as the proportion of patients who achieve complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 during protocol treatment (up to maximum of 6 cycles of treatment) among treated patients.
Duration of response | Up to 1 year
  Will be defined as the time from the date of first documented CR or PR to the date of first documented disease progression or death due to all causes, whichever occurs first.
Progression free survival | Up to 1 year
  Will be defined as the time from the date of registration to the date of first documented disease progression or death due to all causes, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Winston Tan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials